CLINICAL TRIAL: NCT02364726
Title: Acupuncture to Reduce Chemotherapy-induced Peripheral Neuropathy Severity During Neoadjuvant or Adjuvant Weekly Paclitaxel Chemotherapy in Breast Cancer Patients: A Pilot Study
Brief Title: Acupuncture to Reduce Chemotherapy-induced Peripheral Neuropathy Severity During Neoadjuvant or Adjuvant Weekly Paclitaxel Chemotherapy in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-011
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Peripheral Neuropathy
Keywords: Acupuncture; Paclitaxel; 15-011
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Acupuncture Therapy; Surveys and Questionnaires

ARMS (1):
- Acupuncture (Experimental): As part of routine clinical care, a chemotherapy nurse, research nurse, or physician will assess the patient's symptoms including CIPN based on the NCI-CTC 4.0 criteria to determine the grade of CIPN. Once these patients develop National Cancer Institute-Common Toxicity Criteria (NCI-CTC) grade 2 CIPN, they will be recruited for the intervention phase of the study. Severity of CIPN as defined by NCI-CTC is listed in Appendix A. Patients who consent to the intervention phase of the study will then be treated with weekly acupuncture until the end of chemotherapy. No concomitant anti-neuropathy medication will be permitted.
  Subjects will receive acupuncture in bilateral ear points: shen men, point zero, two additional auricular acupuncture point where electrodermal signal is detected and bilateral body acupuncture points: LI4, TE5, LI11, ST40, Ba Feng, Ba xie.
  Interventions: Procedure: Acupuncture; Behavioral: Neuropathic Pain Scale (NPS) questionnaire; Behavioral: FACT/GOG-Ntx questionnaire

INTERVENTIONS:
Procedure: Acupuncture — Each treatment session will be approximately 40 minutes in duration, 10 minutes to insert needles, 30 minutes to leave needles in. Patients will receive one acupuncture treatment each week until the end of chemotherapy. Adverse effects related to the administration of acupuncture will be collected each week before and after each treatment by the acupuncturist or research study assistant. All Integrative Medicine Service acupuncturists are licensed, credentialed employees of MSK.
Behavioral: Neuropathic Pain Scale (NPS) questionnaire — It will be collected weekly throughout the screening phase, as well as, at the time of intervention consent, weekly during the intervention, and then once again after the last acupuncture session before the last chemotherapy session.
Behavioral: FACT/GOG-Ntx questionnaire — It will be collected weekly throughout the screening phase, as well as, at the time of intervention consent, weekly during the intervention, and then once again after the last acupuncture session but before the as the last chemotherapy session, and then once again 3 months (+/-2 weeks) after chemotherapy completion.

SUMMARY:
The purpose of this study is to find out the effects of acupuncture on reducing nerve damage.

Acupuncture is a medical technique of inserting very thin needles into the "energy points" on the body with the aim to restore health and well-being. It has been used widely to treat pain, such as lower back pain and joint pain. In this study the investigators will assess if acupuncture can be used to ease the pain, tingling and numbness that may be caused by chemotherapy and improve quality of life during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Screening Phase:

* Age 21 or older.
* Histologically proven stage I-III carcinoma of the breast.
* Plan to receive adjuvant or neoadjuvant chemotherapy that includes weekly paclitaxel.
* Eastern Cooperative Oncology Group performance status 0-2 (see Appendix B).
* The patient is aware of the nature of his/her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.
* Proficiency in English with the ability to speak and read English.

Exclusion Criteria:

* Known metastatic (stage IV) breast cancer involvement.
* Pre-existing peripheral neuropathy within 28 days of screening consent
* Currently taking anti-neuropathy medication such as gabapentin, pregabalin, duloxetine, or glutamine.

Intervention Phase:

* Age 21 or older.
* Histologically proven stage I-III carcinoma of the breast.
* Receiving adjuvant or neoadjuvant chemotherapy that includes a taxane.
* Eastern Cooperative Oncology Group performance status 0-2
* The patient is aware of the nature of his/her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.
* Proficiency in English with the ability to speak and read English
* While on neurotoxic chemotherapy, has developed NCI-CTC grade 2 CIPN

Exclusion Criteria:

* Known metastatic (stage IV) breast cancer involvement.
* Pre-existing peripheral neuropathy within 28 days of screening consent.
* Currently taking anti-neuropathy medication such as gabapentin, pregabalin, duloxetine, or glutamine.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
CIPN severity as measured by National Cancer Institute-Common Toxicity Criteria version 4.0 | 1 year
  After the initiation of acupuncture through the end of chemotherapy in breast cancer patients undergoing neoadjuvant or adjuvant weekly paclitaxel chemotherapy when compared to historical control ECOG study 1199 [1] weekly paclitaxel treatment arm. The efficacy of acupuncture in reducing CIPN severity and preventing progression of grade 2 CIPN to grade 3 or higher.

SECONDARY OUTCOMES:
CIPN severity as measured by FACT/GOG-Nts | 2 years
  Validated patient-reported outcome questionnaires: Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) questionnaire, the Neuropathy Pain Scale (NPS) and the vibration sensation test will be assessed at the time of intervention consent and then after the last acupuncture session on the same day of the last chemotherapy. CIPN grade per NCI-CTC 4.0 will be assessed weekly and then once again at 3 months (+/-2 weeks) after chemotherapy completion .

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, DABMA, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT02364726/ICF_000.pdf